CLINICAL TRIAL: NCT06056544
Title: A Randomized Clinical Trial of Client-centered Care Coordination to Improve Preexposure Prophylaxis Use for Black Men Who Have Sex With Men
Brief Title: Client-Centered Care Coordination for Black Men Who Have Sex With Men
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Yale University (Other); George Washington University (Other); Us Helping Us, People Into Living, Inc. (Other)
Responsible Party: Principal Investigator, Darren L Whitfield, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HP-00106408; 1R01MH134721 (NIH)
Record Dates: First submitted 2023-09-05; First posted 2023-09-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: HIV Prevention; HIV Pre-exposure Prophylaxis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): C4 is a longitudinal intervention which provides individualized client-centered HIV prevention and support services designed to address health and psychosocial needs that impact the success of PrEP use and adherence (i.e., co-morbidities, substance use, mental health, housing, etc.).
  Interventions: Behavioral: Client Centered Care Coordination
- Control Group (No Intervention): Individuals in the control group will receive standard of care for PrEP use at each clinic. The standard of care is PrEP clinical care includes identifying and engaging patients in need of PrEP, conducting necessary exams and lab tests and prescribing PrEP for the patients, as well as ongoing patient monitoring with follow-up visits and prescriptions-for as long as the patient needs PrEP.

INTERVENTIONS:
Behavioral: Client Centered Care Coordination — During the initial C4 sessions, participants will be offered PrEP. For participants who initiate PrEP, C4 staff will provide an individualized PrEP initiation plan. During subsequent C4 sessions, C4 staff will review the prevention plan and goals with participants and use autonomy supportive counseling to address the barriers that are identified by participants that impact their motivation to use PrEP and adhere to PrEP through referrals to support services (e.g, PrEP access programs, addiction medicine services, housing, and job resources). In addition, the C4 staff will ensure any medical issues related to PrEP adherence are addressed by the site medical providers.
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to determine the efficacy of a client-center care coordination intervention (C4) in improving pre-exposure prophylaxis (PrEP) adherence in Black men who have sex with men (MSM). The main aims of the study are:

1. Determine the efficacy of C4 for increasing PrEP adherence among Black MSM.
2. Identify the optimal dose of C4 implementation for maximizing its effect on PrEP adherence.
3. Describe the acceptability and feasibility of C4 implementation in community settings.

Participants in the clinical trial will be randomized to receive the intervention or standard of care for PrEP in two sites. Researchers will compare administration of C4 to standard of care to see if C4 improves adherence to PrEP. C4 is a longitudinal intervention which provides individualized client-centered HIV prevention and support services designed to address health and psychosocial needs that impact the success of PrEP use and adherence (i.e., co-morbidities, substance use, mental health, housing, etc.). The intervention pulls from the Centers for Disease Control and Prevention (CDC) Comprehensive Risk Counseling and Services (CRCS) and Self-Determination Theory (SDT) to support client-identified HIV prevention goals to promote, adopt, and maintain PrEP use. CRCS is a public health strategy to assist persons in developing behavioral goals to reduce HIV acquisition and transmission. In this intervention, the HIV prevention plan element of CRCS will be the foundation of the C4 intervention. After the initial prevention plan is developed, elements of SDT will be used to implement a client-centered care approach to assist in addressing issues which many arise which impede successful PrEP adherence.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years of age
* Identify as Black, African American, Black African, Afro-Caribbean, or Black-Latino
* Cisgender male
* PrEP naïve or who prematurely stopped PrEP
* No prior HIV diagnosis confirmed through HIV testing
* Self-reported high risk for acquiring HIV
* Currently not enrolled in another HIV prevention study

Exclusion Criteria:

* Black MSM who received a reactive or positive HIV test at screening or self report HIV-positive
* Identifying as transgender
* Current participation in any research study via self-report
* Use of PrEP or post-exposure prophylaxis in the last 60 days prior to anticipated enrollment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
PrEP Adherence | 6, 12, 18 months
  Count of doses of PrEP missed in the last 30 days by self report
PrEP Adherence | 6, 12, 18 months
  Number of participants with tenofovir-diphosphate (fmol/punch) of greater than 700 using dried blood spots analyzing peripheral blood mononuclear cells (PBMCs) and plasma concentration assay for tenofovir-diphosphate (TFV-DF) and emtricitabine-triphosphate (FTC-TP).

CONTACTS AND LOCATIONS:
Locations (1):
- Us Helping Us, People Into Living Inc., Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing ensures the ability of translation of research results into knowledge, research products, and interventions to improve the health of communities. The research team commits to transparency through sharing the data generated by this project. All research data will be shared as requested in accordance with federal regulations and the Freedom of Information Act. The research team anticipates dissemination of results beginning in the 4th year of the award period. Sharing of the findings will involve a primary paper describing the effectiveness of the intervention on pre-exposure prophylaxis (PrEP) use and adherence and secondary papers reporting the qualitative findings and sub-analyses. Study findings will also be shared in the form of scientific and community presentations.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The final study data set will be shared through Inter-university Consortium for Political and Social Research (ICPSR) no later than the time of acceptance of the secondary paper on the qualitative findings on feasibility and acceptability of the intervention. Based on our study timeline, we expect this to be approximately spring of 2029, although the actual date could be earlier or later depending on the time for completing data analysis.